CLINICAL TRIAL: NCT02607553
Title: G-202-006: An Open-Label, Single-Arm, Phase II Study to Evaluate the Safety and Activity of G-202 in Patients With Clear Cell Renal Cell Carcinoma That Expresses PSMA
Brief Title: Safety and Activity of G-202 in Patients With Clear Cell Renal Cell Carcinoma That Expresses PSMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-006
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: G-202 (Experimental): G-202 administered by intravenous infusion on 3 consecutive days of a 28-day cycle
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — G-202 administered by intravenous infusion on Days 1, 2 and 3 of each 28-day cycle until disease progression
  Other Names: Mipsagargin

SUMMARY:
An open-label, single-arm, single-center Phase II study to evaluate the safety and activity of G-202 in patients with clear cell renal cell carcinoma that expresses PSMA

DETAILED DESCRIPTION:
Epithelial tumors, including clear cell renal cell carcinoma (RCC), have the ability to grow to only a finite size in the absence of vascularization. RCC is characterized as a highly-vascularized tumor and inhibiting angiogenesis has the potential to impair tumor growth, including growth of RCC. Therapeutic targeting of integral biological pathways in RCC, including those involving VEGF and mTOR, has produced robust clinical effects and revolutionized the treatment of metastatic RCC. These approaches offers significant clinical benefit and sequential use of these agents has become the empirical standard of care. However, complete or durable responses are uncommon and resistance develops after a median interval of 6-15 months. This raises the pressing clinical need for additional therapeutic approaches for patients with metastatic clear cell RCC. The purpose of this study is to investigate the approach of targeted delivery of cytotoxic chemotherapy with G-202 in patients with advanced, refractory RCC. This study is based on prodrug tumor targeting, in which an inactive form of a toxic agent is administered systemically and gets activated in specific locations in the body, resulting in higher concentrations of the cytotoxic form at the tumor location. G-202 is a prodrug that is activated by PSMA in the blood vessels of tumors, but not normal tissue; once activated, G-202 leads to disruption of intracellular calcium levels and subsequent induction of apoptosis. Thus, G-202 is expected to bring about cell death in RCC and destroy the blood supply of RCC tumors. This single-arm, open-label Phase II clinical trial will evaluate the safety and activity of G-202 in patients with RCC that expresses PSMA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥ 18 years
* Pathologic documentation of clear cell renal cell carcinoma
* Disease that is resistant or refractory to standard of care
* ECOG Performance Status < 2
* Most recent tissue biopsy demonstrates PSMA expression by immunohistochemical staining
* Adequate bone marrow function measured within 7 days prior to first infusion of G-202 (absolute peripheral granulocyte count > 1500 cells/m3; platelet count > 100,000 cells/m3)
* Adequate hepatic function measured within 7 days prior to first infusion of G-202 (Albumin ≥ 2.8 g/dL; AST and ALT ≤ 5 x ULN; Total bilirubin <2 mg/dL)
* Adequate renal function measured within 7 days prior to first infusion of G-202 (Proteinuria level ≤ 2 by urine dipstick; Serum creatinine ≤1.5 x ULN)
* Normal coagulation profile measured within 14 days prior to first infusion of G-202 (INR ≤ 2.3; aPTT ≤ 1.5 X ULN)
* No history of substantial non-iatrogenic bleeding diatheses. Use of anti-coagulants is limited to local use only (for control of central line patency)
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study and are willing to participate in the study
* Females of child-bearing potential and males with female partners of child-bearing potential must be willing to use acceptable methods of contraception to avoid pregnancy (for example, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) beginning before the first infusion of G-202 and for 3 months after the last infusion of G-202

Exclusion Criteria:

* Uncontrolled cardiac, hepatic, renal, or neurologic/psychiatric disorder
* HIV positivity or history of chronic hepatitis B or C infection
* Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, unless a 2D echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months of enrollment demonstrates a left ventricular ejection fraction >45%
* History of another malignancy within the previous 5 years other than curatively treated non-melanoma skin cancer or or intraepithelial carcinoma of the cervix
* Surgical resection or major surgery within 4 weeks or stereotactic biopsy within 1 week of first G-202 treatment
* Treatment, chemotherapy, radiation therapy, immunotherapy, or investigational drug for the patient's renal cell cancer within 28 days prior to first infusion of G-202
* Currently requiring systemic administration of antibiotics or chronic administration of anti-viral agents
* Use of anti-coagulants is limited to local use for control of central line patency
* History or evidence of cardiac risk, including corrected QT interval on screening ECG > 470 msec, clinically significant uncontrolled arrhythmias or arrhythmia requiring treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia, history of acute coronary syndromes within 6 months prior to the first dose of study therapy (including myocardial infarction and unstable angina, coronary artery bypass graft, angioplasty, or stenting), any history of congestive heart failure with most recent ejection fraction < 45%
* Uncontrolled cardiac or coronary artery disease
* Uncontrolled hypertension (mean systolic BP ≥ 160 mm Hg and/or mean diastolic BP ≥ 100 mm Hg on 3 determinations 5 minutes apart while on 2 anti-hypertensive agents) or hypertension requiring treatment with more than 2 anti-hypertensive agents.
* Severe or uncontrolled medical disease, including uncontrolled diabetes, congestive heart failure, chronic renal disease or chronic pulmonary disease
* Severe gastrointestinal bleeding within 12 weeks of treatment with G-202
* Requirement for chronic use of medications known to be strong inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes (Appendix 3) Note: If patients can stop receiving these medications, CYP3A4 inhibitors should be discontinued at least 7 days prior to starting treatment with G-202
* Known hypersensitivity to any study drug component including thapsigargin derivatives, polysorbate 20, or propylene glycol
* Any other condition, including concurrent medical condition, social circumstance or drug dependency, which in the opinion of the investigator could compromise patient safety and/or compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Clinical activity | 8 weeks from first administration of G-202
  Use RECIST criteria to assess the clinical activity of G-202 administered by intravenous infusion daily for 3 consecutive days of a 28-day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Robert Amato, D.O., Principal Investigator — University of Texas Health Sciences Center at Houston
Locations (1):
- University of Texas Health Science Center, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No